CLINICAL TRIAL: NCT05232539
Title: Efficiency of Intraoperative Optical Coherence Tomography (iOCT) in Eye Surgery
Brief Title: Efficiency of Intraoperative Optical Coherence Tomography (iOCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Somich, s.r.o. (Other)
Collaborators: Vascular surgery, University hospital Královské Vinohrady, Prague (Other)
Responsible Party: Principal Investigator, Tomas Benda, MD, FEBO, Principal Investigator, Somich, s.r.o.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IOCT2022
Record Dates: First submitted 2022-01-15; First posted 2022-02-10 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Epiretinal Membrane; Glaucoma; Cornea
Keywords: Intraoperative OCT
MeSH Terms: conditions — Epiretinal Membrane; Glaucoma; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, comparative study conducted at the SOMICH Eye Center s.r.o. in Karlovy Vary, comparing the effectiveness and safety of the use of Intraoperative Optical Coherence Tomography (iOCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Lamellar corneal transplantation type DMEK (Active Comparator): 50 operations, procedure will be randomly divided into 2 subgroups of 25 patients with and without the use of iOCT during the operation.
  Interventions: Device: Intraoperative Optical Coherence Tomography (iOCT)
- Deep sclerectomy with implantation of subchoroidal implant Esnoper Clip (Active Comparator): 50 operations, procedure will be randomly divided into 2 subgroups of 25 patients with and without the use of iOCT during the operation.
  Interventions: Device: Intraoperative Optical Coherence Tomography (iOCT)
- Pars plana vitrectomy with epiretinal membrane peeling (Active Comparator): 50 operations, procedure will be randomly divided into 2 subgroups of 25 patients with and without the use of iOCT during the operation.
  Interventions: Device: Intraoperative Optical Coherence Tomography (iOCT)

INTERVENTIONS:
Device: Intraoperative Optical Coherence Tomography (iOCT) — The use of iOCT during surgery offers the advantage of a new view of the operating field, theoretically allows more precise performance and can also change decision-making mechanisms during surgery with more precise visual control of some surgical steps.

SUMMARY:
Efficiency of Intraoperative Optical Coherence Tomography (iOCT)

Hypothesis:

The use of iOCT during surgery offers the advantage of a new view of the operating field, theoretically allows more precise performance and can also change decision-making mechanisms during surgery with more precise visual control of some surgical steps (incision adaptation, differentiation of healthy and pathological tissue, placement of the implant, graft, etc.) The disadvantage is the prolongation of the operation and thus the theoretical increase in possible complications related to the operation (bleeding, infection, patient subjective problems - pain, restlessness, poorer cooperation and the resulting other possible risks, such as unexpected patient movement).

Aim:

Determining the effectiveness of iOCT use in different types of eye surgery. Evaluation of advantages and disadvantages of using iOCT.

DETAILED DESCRIPTION:
Methods:

The effectiveness of iOCT use will be monitored in three types of microsurgical eye surgery:

1. Lamellar corneal transplantation type DMEK
2. Antiglaucoma surgery - Deep sclerectomy with implantation of subchoroidal implant Esnoper Clip
3. Pars plana vitrectomy with epiretinal membrane peeling

For each type of the surgery, the investigators expect to perform about 50 surgeries, individual procedures will be randomly divided into 2 subgroups of 25 patients with and without the use of iOCT during the operation.

Perioperatively, the surgeon will record the number of complications, the net time of the operation and impressions using a questionnaire. The patient will evaluate the subjective perception of the operation using a questionnaire (pain, pressure, subjectively perceived duration of the operation).

The investigators will evaluate the clinical outcome of the operation postoperatively at intervals of 1 week, 1, 3 and 6 months - corrected and uncorrected visual acuity, intraocular pressure, inflammation reaction (SUN - standardization of uveitis nomenclature) and possible postoperative complications in all groups.

In each group the investigators will also specifically evaluate the achievement of the planned surgical goal in the group:

1. attachment of the lamella (respectively% area of lamella ablation) on the slit lamp, number of necessary reoperations - rebubbling, and density of the transplanted endothelium using the endothelial microscope
2. correct localization of the Esnoper Clip implant and confirmation of its functionality (decentration of the implant in millimeters, functionality expressed by the size of filtration into the subcleral and suprachoroidal space (using stationary OCT), the amount of postoperative antiglaucoma therapy required).
3. Frequency of epiretinal membrane residues (using stationary OCT)
4. Histological verification of tissues identified on the basis of iOCT during surgery (in Deep sclerectomy and Pars plana vitrectomy patients)

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Bullous keratopathy and Fuchs dystrophy of the cornea indicated for surgical treatment DMEK
2. Clinical diagnosis of Primary open angle glaucoma and Normotension glaucoma indicated for surgical treatment Deep sclerectomy with implantation of subchoroidal implant Esnoper Clip
3. Clinical diagnosis of Epiretinal membrane indicated for surgical treatment Pars plana vitrectomy with epiretinal membrane peeling

Exclusion Criteria:

1. If it is not possible to take an iOCT image
2. Uveitis in anamnestic history
3. Other ocular diagnosis deteriorating visual acuity (eg. age related macular degeneration, diabetic macular edema, macular scars)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Attachment of the transplanted DMEK lamella. | At the first week postoperatively.
  The investigators will evaluate the attachment of the transplanted DMEK lamella (respectively % area of lamella ablation) on the slit lamp.
Attachment of the transplanted DMEK lamella. | 1 month postoperatively
  The investigators will evaluate the attachment of the transplanted DMEK lamella (respectively % area of lamella ablation) on the slit lamp.
Attachment of the transplanted DMEK lamella. | 3 months postoperatively
  The investigators will evaluate the attachment of the transplanted DMEK lamella (respectively % area of lamella ablation) on the slit lamp.
Attachment of the transplanted DMEK lamella. | 6 months postoperatively
  The investigators will evaluate the attachment of the transplanted DMEK lamella (respectively % area of lamella ablation) on the slit lamp.
Density of the transplanted endothelium cells. | At the first week postoperatively.
  The investigators will evaluate the density of the transplanted endothelium cells using the endothelial microscope.
Density of the transplanted endothelium cells. | 1 month postoperatively
  The investigators will evaluate the density of the transplanted endothelium cells using the endothelial microscope.
Density of the transplanted endothelium cells. | 3 months postoperatively
  The investigators will evaluate the density of the transplanted endothelium cells using the endothelial microscope.
Density of the transplanted endothelium cells. | 6 months postoperatively
  The investigators will evaluate the density of the transplanted endothelium cells using the endothelial microscope.
Correct localization of the Esnoper Clip implant and confirmation of its functionality. | At the first week postoperatively.
  The investigators will evaluate correct localization of the Esnoper Clip implant and confirmation of its functionality (decentration of the implant in millimeters, functionality expressed by the size of filtration into the subcleral and suprachoroidal space) using stationary OCT.
Correct localization of the Esnoper Clip implant and confirmation of its functionality. | 1 month postoperatively
  The investigators will evaluate correct localization of the Esnoper Clip implant and confirmation of its functionality (decentration of the implant in millimeters, functionality expressed by the size of filtration into the subcleral and suprachoroidal space) using stationary OCT.
Correct localization of the Esnoper Clip implant and confirmation of its functionality. | 3 months postoperatively
  The investigators will evaluate correct localization of the Esnoper Clip implant and confirmation of its functionality (decentration of the implant in millimeters, functionality expressed by the size of filtration into the subcleral and suprachoroidal space) using stationary OCT.
Correct localization of the Esnoper Clip implant and confirmation of its functionality. | 6 months postoperatively
  The investigators will evaluate correct localization of the Esnoper Clip implant and confirmation of its functionality (decentration of the implant in millimeters, functionality expressed by the size of filtration into the subcleral and suprachoroidal space) using stationary OCT.
Frequency of epiretinal membrane residues. | At the first week postoperatively.
  The investigators will evaluate the frequency of epiretinal membrane residues using stationary OCT.
Histological verification of tissues identified on the basis of iOCT during surgery. | At the first week postoperatively.
  The investigators in cooperation with pathologist will histologicaly verificate tissues identified on the basis of iOCT during surgery in Deep sclerectomy and Pars plana vitrectomy patients.

SECONDARY OUTCOMES:
Inflammation reaction | At the first week postoperatively.
  The investigators will evaluate intraocular postoperative inflammation reaction using the SUN - standardization of uveitis nomenclature
Inflammation reaction | 1 month postoperatively
  The investigators will evaluate intraocular postoperative inflammation reaction using the SUN - standardization of uveitis nomenclature
Inflammation reaction | 3 months postoperatively
  The investigators will evaluate intraocular postoperative inflammation reaction using the SUN - standardization of uveitis nomenclature
Inflammation reaction | 6 months postoperatively
  The investigators will evaluate intraocular postoperative inflammation reaction using the SUN - standardization of uveitis nomenclature
Visual acuity | At the first week postoperatively.
  The investigators will evaluate corrected and uncorrected visual acuity on LogMAR chart.
Visual acuity | 1 month postoperatively
  The investigators will evaluate corrected and uncorrected visual acuity on LogMAR chart.
Visual acuity | 3 months postoperatively
  The investigators will evaluate corrected and uncorrected visual acuity on LogMAR chart.
Visual acuity | 6 months postoperatively
  The investigators will evaluate corrected and uncorrected visual acuity on LogMAR chart.
Intraocular pressure | At the first week postoperatively.
  The investigators will evaluate intraocular pressure using non-contact tonometry in mmHg.
Intraocular pressure | 1 month postoperatively
  The investigators will evaluate intraocular pressure using non-contact tonometry in mmHg.
Intraocular pressure | 3 months postoperatively
  The investigators will evaluate intraocular pressure using non-contact tonometry in mmHg.
Intraocular pressure | 6 months postoperatively
  The investigators will evaluate intraocular pressure using non-contact tonometry in mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Somich, Karlovy Vary, Czechia

IPD SHARING:
Plan to Share IPD: No